CLINICAL TRIAL: NCT05080881
Title: Noninvasive Monitor of Vascular Volume Fluid Shifts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to close the study.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James C. Leiter, Principal Investigator, Professor of Molecular and Systems Biology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D18144
Record Dates: First submitted 2021-09-22; First posted 2021-10-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Blood Loss
Keywords: phonocardiographic measurements
MeSH Terms: conditions — Hemorrhage | interventions — Cardiography, Impedance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood draw (Experimental): All blood draw subjects will have baseline data collected over 15 minutes. The participants with then donate blood. For 15 minutes after the blood donation, the participant will stay in place and will continue to have data collected.
  Interventions: Diagnostic Test: phonocardiographic measurement: InnoVital Systems; Diagnostic Test: phonocardiographic measurement: ThinkLabs StethOne; Diagnostic Test: physiological measurements: BIOPAC; Diagnostic Test: physiological measurements: Masimo Radical-7; Diagnostic Test: physiological measurements: CoVa Monitoring System 2; Diagnostic Test: Thoracic impedance

INTERVENTIONS:
Diagnostic Test: phonocardiographic measurement: InnoVital Systems — The instrument consists of one or more low-profile microphones in plastic housings with nitrile or silicon diaphragms. These sensors convert heart sounds into analog signals that will be acquired by the BIOPAC data acquisition system.
  Other Names: InnoVital Systems
Diagnostic Test: phonocardiographic measurement: ThinkLabs StethOne — This device senses heart sounds and may be listened to using headphones and converted to an analog signal and saved using the BIOPAC data acquisition system.
  Other Names: ThinkLabs StethOne
Diagnostic Test: physiological measurements: BIOPAC — Non-invasive blood pressure, electrocardiogram, heart rate, respiratory rate, and leg circumference - This is a commercially available device used regularly in health care settings to monitor continual blood pressure and heart rate.
  Other Names: BIOPAC
Diagnostic Test: physiological measurements: Masimo Radical-7 — A commercially available device for pulse oximetry and continuous non-invasive hematocrit measurement.
  Other Names: Masimo Radical-7
Diagnostic Test: physiological measurements: CoVa Monitoring System 2 — This device will be used for thoracic bioimpedance and other physiological measures. This is a commercially available device. It also measures ECG, heart rate, heart rate variability, estimated stroke volume, and estimated cardiac output. The study team may measure either while body bioimpedance or thoracic bioimpedance.
  Other Names: CoVa Monitoring System 2
Diagnostic Test: Thoracic impedance — Thoracic impedance is measured using the Starling device (https://usstarling.baxter.com/starling-system). Baxter uses a series of proprietary algorithms to infer stroke volume and cardiac output from thoracis impedance. Calculated values will be recorded, but the main variable that will be recorded is simply the temporal profile of thoracic impedance during the manipulations in each group (changing lower body negative pressure or therapeutic phlebotomy).
  Other Names: Baxter

SUMMARY:
Blood volume measurements are a critical step in the emergency care of trauma patients. The typical approach to this is to rely on historical information, physical examination and metrics such as heart rate. There is currently no good real-time measure to track blood volume. This study investigates the use of phonocardiography (listening to the sounds made by the heart) to track changes in central blood volume.

DETAILED DESCRIPTION:
Blood draw subjects:

Participation in this study group may last up to 60 minutes. Participants will begin with a brief medical exam to determine eligibility. This will include a review of any history of cardiovascular disease and of medications. Prior to a scheduled blood draw, eligible participates will have physiological measurements taken, which may include phonocardiographic measurements, cardiac output, plethysmography (volume changes), multifrequency bioimpedance, thoracic impedance, heart rate, blood pressure, pulse oximetry, continuous non-invasive hematocrit measurement, and respiration. The phonocardiographic measurements may be taken with both a commercial and a custom-built device. These are all non-invasive measurements. After 15 minutes of baseline measurements, a blood draw will proceed normally while the physiological measurements continue. After the participant is finished donating blood, the participant will be asked to stay in place for an additional 15 minutes to continue to collect physiological data. Participants are asked not to eat or drink during the 15 minutes as this will provide better data collection. The information collected as data for this study includes: information about medical history, body measurements, and physiological measurements.

ELIGIBILITY:
Lower Body Negative Pressure (LBNP) participants:

Inclusion Criteria:

* In generally good health
* Free of systemic diseases
* No contraindications to LBNP exposure.
* No prior history of cardiovascular disease
* Normal resting systolic blood pressure (SBP, 100-140 mm Hg) and diastolic blood pressure (DBP, 60-90 mm Hg).

Exclusion Criteria:

* Individuals who, after lying supine for five minutes, show a greater than 10 mm Hg drop in systolic pressure or a greater than 20 beats/minute increase in heart rate with standing during pre-enrollment evaluation

Blood draw participants:

Inclusion Criteria:

* In generally good health
* Free of systemic diseases
* No current or prior history of cardiovascular disease or cardiovascular reactive drugs
* Blood donors through the DHMC blood donation center
* Healthy volunteers
* People who are taking part in another study where about 500 ml of blood is being drawn
* Therapeutic phlebotomy patients (hemochromatosis or polycythemia vera patients)

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in cardiac cycle time intervals | Through study completion; 3 hours
  Cardiac systolic and diastolic times
Change in phonographic characteristics - amplitude | Through study completion; 3 hours
  Size of cardiac systolic and diastolic heart tones
Change in phonographic characteristics - frequency | Through study completion; 3 hours
  Frequency content of cardiac tones

CONTACTS AND LOCATIONS:
Overall Officials: James C Leiter, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are no data to share.